CLINICAL TRIAL: NCT03047993
Title: Phase Ib/II Study of the Glutaminase Inhibitor CB-839 in Combination With Azacitidine in Patients With Advanced Myelodysplastic Syndrome
Brief Title: Glutaminase Inhibitor CB-839 and Azacitidine in Treating Patients With Advanced Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0636; NCI-2018-01243 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0636 (Other: M D Anderson Cancer Center); R01CA206210 (NIH)
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia; Blasts 20-30 Percent of Bone Marrow Nucleated Cells; Blasts 20-30 Percent of Peripheral Blood White Cells; Chronic Myelomonocytic Leukemia; High Risk Myelodysplastic Syndrome; IPSS Risk Category Intermediate-2; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Azacitidine; CB-839

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (glutaminase inhibitor CB-839, azacitidine) (Experimental): Patients receive glutaminase inhibitor CB-839 PO BID on days 1-28 and azacitidine SC or IV over 10-40 minutes on days 1-7.
  Interventions: Drug: Azacitidine; Drug: Glutaminase Inhibitor CB-839

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Glutaminase Inhibitor CB-839 — Given PO
  Other Names: CB-839

SUMMARY:
This phase I/II trial studies the side effects of glutaminase inhibitor CB-839 in combination with azacitidine in treating patients with myelodysplastic syndrome that has spread to other places in the body. Glutaminase inhibitor CB-839 and azacitidine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability and clinical activity of glutaminase inhibitor CB-839 (CB-839) in combination with azacitidine (AZA) for patients with advanced myelodysplastic syndrome (MDS).

SECONDARY OBJECTIVES:

I. To explore the pharmacokinetics (PK) of CB-839 in combination with AZA. II. To explore the pharmacodynamics (PDn) of CB-839 in combination with AZA. III. To assess overall survival, event-free survival and duration of response of CB-839 in combination with AZA.

OUTLINE:

Patients receive glutaminase inhibitor CB-839 orally (PO) twice daily (BID) on days 1-28 and azacitidine subcutaneously (SC) or intravenously (IV) over 10-40 minutes on days 1-7.

After completion of study treatment, patients are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent must be obtained prior to any study specific procedures
* Subjects with a histologically confirmed diagnosis of MDS, including both MDS and refractory anemia with excess blasts (RAEB)-T (acute myeloid leukemia [AML] with 20-30% blasts and multilineage dysplasia by French-American-British [FAB] criteria) by World Health Organization (WHO) and chronic myelomonocytic leukemia (CMML) are eligible
* Subjects with high-risk MDS (i.e. International Prognostic Scoring System [IPSS] Intermediate-2 or high-risk; or R-IPSS high or very-high risk). Patients with Intermediate-1 risk by IPSS or Intermediate risk by R-IPSS and with IDH1 or IDH2, or high-risk molecular features including TP53, ASXL1, EZH2, and/or RUNX1 mutations are also eligible
* Subjects with prior hypomethylating agent therapy exposure may be eligible based on discussion with the principal investigator (PI)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Serum bilirubin =< 2 x the upper limit of normal (ULN) (except for patients with Gilbert's disease)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 3 x the laboratory ULN
* Creatinine clearance > 30 mL/min based on the Cockcroft-Gault equation
* Able to understand and voluntarily sign a written informed consent, and willing and able to comply with protocol requirements
* Resolution of all treatment-related, non-hematological toxicities, except alopecia, from any previous cancer therapy to < grade 1 prior to the first dose of study treatment
* Female patients of childbearing potential must have a negative serum or urine pregnancy test within 3 days of the first dose of study drug and agree to use dual methods of contraception during the study and for a minimum of 3 months following the last dose of study drug. Post-menopausal females (>= 45 years old and without menses for >= 1 year) and surgically sterilized females are exempt from these requirements. Male patients must use an effective barrier method of contraception during the study and for a minimum of 3 months following the last dose of study drug if sexually active with a female of childbearing potential

Exclusion Criteria:

* Any prior or coexisting medical condition that in the investigator's judgment will substantially increase the risk associated with the subject's participation in the study
* Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures
* Active uncontrolled infection at study enrollment including known diagnosis of human immunodeficiency virus or chronic active hepatitis B or C infection
* Clinically significant gastrointestinal conditions or disorders that may interfere with study drug absorption, including prior gastrectomy
* Patients with known active central nervous system (CNS) disease, including leptomeningeal involvement
* Impaired cardiac function, uncontrolled cardiac arrhythmia, or clinically significant cardiac disease including the following: a) New York Heart Association grade III or IV congestive heart failure, b) myocardial infarction within the last 6 months
* Subjects with a corrected QT (QTc) > 480 ms (QTc > 510 msec for subjects with a bundle branch block at baseline)
* Nursing or pregnant women
* Subjects with known hypersensitivity to study drugs or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] DiNardo CD, Verma D, Baran N, Bhagat TD, Skwarska A, Lodi A, Saxena K, Cai T, Su X, Guerra VA, Poigaialwar G, Kuruvilla VM, Konoplev S, Gordon-Mitchell S, Pradhan K, Aluri S, Hackman GL, Chaudhry S, Collins M, Sweeney SR, Busquets J, Rathore AS, Deng Q, Green MR, Grant S, Demo S, Choudhary GS, Sahu S, Agarwal B, Spodek M, Thiruthuvanathan V, Will B, Steidl U, Tippett GD, Burger J, Borthakur G, Jabbour E, Pemmaraju N, Kadia T, Kornblau S, Daver NG, Naqvi K, Short NJ, Garcia-Manero G, Tiziani S, Verma A, Konopleva M. Glutaminase inhibition in combination with azacytidine in myelodysplastic syndromes: a phase 1b/2 clinical trial and correlative analyses. Nat Cancer. 2024 Oct;5(10):1515-1533. doi: 10.1038/s43018-024-00811-3. Epub 2024 Sep 19. PMID 39300320
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Glutaminase Inhibitor CB-839, Azacitidine)
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Glutaminase Inhibitor CB-839, Azacitidine)
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 70 [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Response is Complete Remission (CR) + Partial Remission (PR) + Marrow CR = Complete Remission (CR) is </=5% myeloblasts with normal maturation of all cell lines* Persistent dysplasia will be noted, Peripheral blood; hemoglobin>/=11 g/dL, Platelets >/= 100x10^9/L ,Neutrophils >/=1.0 x 10^9/L, Blasts = 0%. Partial Remission (PR) is all CR criteria if abnormal before treatment except: Bone marrow blasts decreased by </=50% over pretreatment but still >5% Cellularity and morphology not relevant. Marrow CR is Bone marrow: </= 5% meyloblasts and decreased by >/= 50% over pretreatment† Peripheral blood: if HI responses, they will be noted in addition to marrow CR.
Time Frame: Up to 5 years, 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glutaminase Inhibitor CB-839, Azacitidine)
Number analyzed (Participants) | 28
Participants | 11

ADVERSE EVENTS:
Time Frame: Up to 5 years, 4 months
Arm/Group | Treatment (Glutaminase Inhibitor CB-839, Azacitidine)
All-Cause Mortality (participants affected / at risk) | 6/28
Serious Adverse Events (participants affected / at risk) | 18/28
Other Adverse Events (participants affected / at risk) | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Glutaminase Inhibitor CB-839, Azacitidine) (N=28)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Blood and lymphatic disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Cardiac Disorders, Other - Decompensated Heart Failure (Cardiac disorders) | 2 (2)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal Disorders, Other-Melena (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Disorders-Hemorrhage (Gastrointestinal disorders) | 1 (2)
General disorders and administration site conditions-Other, Neck Swelling (General disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Immune System Disorders, Other (Immune system disorders) | 1 (1)
Infection (Infections and infestations) | 4 (5)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Lung infection (Infections and infestations) | 2 (2)
Mucositis (Gastrointestinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1)
Soft tissue Infection (Infections and infestations) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Vascular Disorders, Other-Hematoma (Vascular disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Death (General disorders) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT03047993/Prot_SAP_001.pdf